CLINICAL TRIAL: NCT02501902
Title: AN OPEN-LABEL PHASE IB STUDY OF PALBOCICLIB (ORAL CDK 4/6 INHIBITOR) PLUS ABRAXANE (REGISTERED) (NAB-PACLITAXEL) IN PATIENTS WITH METASTATIC PANCREATIC DUCTAL ADENOCARCINOMA
Brief Title: Dose-Escalation Study Of Palbociclib + Nab-Paclitaxel In mPDAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A5481059; 2015-001307-31 (EudraCT Number)
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Ibrance, palbociclib, Abraxane, nab-paclitaxel, pancreas,
MeSH Terms: interventions — palbociclib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palbociclib + Nab-Paclitaxel (Experimental): Palbociclib oral dosing on Days 1 to 21 of each 28-day cycle. Nab-paclitaxel IV dosing on Days -2, 6, and 13 of Cycle 1, and on Days 1, 8, and 15 of subsequent cycles.
  Interventions: Drug: Palbociclib; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Palbociclib — Palbociclib oral dosing on Days 1 to 21 of each 28-day cycle.
  Other Names: Ibrance
Drug: Nab-Paclitaxel — Nab-paclitaxel IV dosing on Days -2, 6, and 13 of Cycle 1, and on Days 1, 8, and 15 of subsequent cycles.
  Other Names: Abraxane

SUMMARY:
This is a Phase 1, open label, multi center, multiple dose, dose escalation, safety, pharmacokinetic and pharmacodynamic study of palbociclib in combination with nab-P, in sequential cohorts of adult patients with mPDAC, with MTD expansion cohort(s). Approximately 30-60 patients are expected to be enrolled in the overall study.

DETAILED DESCRIPTION:
The study has 2 parts:

• Part A (Dose-Escalation Cohorts): Consecutive cohorts of patients will receive escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles, in order to estimate the MTD(s) of the combination. The starting doses will be 75 mg palbociclib, and 100 mg/m2 nab-P. The observation period for dose-limiting toxicities (DLTs) will be from Day 1 to Day 28. Pharmacokinetic (PK) and pharmacodynamic (PD) properties of palbociclib and nab-P will also be assessed. Up to approximately 30 patients will be enrolled. The criteria for dose escalation will be based on a modified toxicity probability interval (mTPI) method.

• Part B [MTD Expansion Cohort(s)]: When the MTD(s) of palbociclib plus nab-P has been estimated with confidence, enrollment will proceed into 1 or 2 MTD expansion cohort(s) of up to 20 patients each at the MTD(s). The objective of the MTD expansion cohort(s) will be to provide additional information on safety, tolerability, biomarkers, PD activity, and PK/PD relationship for the combination regimen in order to determine the RP2D. The MTD expansion cohort(s) will only enroll patients who have not received previous treatment for their metastatic disease in order to evaluate preliminary activity of the combination in the target patient population.

All patients (in Part A and B) will receive nab-P intravenously once weekly for 3 weeks out of each 28-day cycle. Palbociclib oral dosing will be once daily on Days 1-21 of each 28-day cycle. To allow for PK evaluation of nab-P administered alone, nab-P will be administered on Day -2 for Cycle 1 only. Subsequent cycles will administer both nab-P and palbociclib on Day 1. Alternate dosing schedules for palbociclib may be explored based on emerging PK, PD, and safety data.

Patients will be treated as long as they are clinically benefiting from investigational product without unacceptable toxicity, objective disease progression, or withdrawal of consent. A modified visit schedule will be implemented for patients who are on investigational product for more than 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed metastatic pancreatic ductal adenocarcinoma.
* Availability of a tumor tissue specimen. If no archived tumor tissue is available, then a de novo biopsy is required for patient participation.
* Karnofsky Performance Status 70 or greater.
* Adequate Bone Marrow, Renal, and Liver Function.

Exclusion Criteria:

* Prior treatment with a CDK 4/6 inhibitor.
* Prior treatment with nab-P for the treatment of metastatic disease.
* Patients with known CNS metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth.
* Diagnosis of any other malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* QTc >480 msec, or family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes.
* Uncontrolled electrolyte disorders.
* Cardiac or pulmonary disorders within 6 months of enrollment.
* Known human immunodeficiency virus infection.
* History of interstitial lung disease or pneumonitis.
* Other severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nab-P.
* Difficulty swallowing capsules or requirement for a feeding tube.
* Previous high-dose chemotherapy requiring stem cell rescue.
* Pregnant female patients; breastfeeding female patients; male patients with partners currently pregnant.
* Active inflammatory or other gastrointestinal disease,
* Active bleeding disorder in the past 6 months.
* Patients treated within the last 7 days prior to the start of IP with strong/moderate CYP3A4 inhibitors, strong/moderate CYP3A4 inducers, CYP2C8 inhibitors, strong/moderate CYP2C8 inducers, or drugs that are known to prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (21):
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - Virginia G. Piper Cancer Pharmacy, Scottsdale, Arizona
  - UC San Diego Medical Center - La Jolla (Thornton Hospital), La Jolla, California
  - UC San Diego Moores Cancer Center - Investigational Drug Services, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Denver, CTO (CTRC), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
- Spain (5):
  - Hospital Universitario de Fuenlabrada. Unidad de Farmacia, Fuenlabrada, Madrid
  - Hospital Universitario Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitari Vall D'Hebron, Servicio de Oncología Médica, Barcelona
  - Hospital Universitario 12 de Octubre Servicio de Farmacia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Hidalgo M, Garcia-Carbonero R, Lim KH, Messersmith WA, Garrido-Laguna I, Borazanci E, Lowy AM, Medina Rodriguez L, Laheru D, Salvador-Barbero B, Malumbres M, Shields DJ, Grossman JE, Huang X, Tammaro M, Martini JF, Yu Y, Kern K, Macarulla T. A Preclinical and Phase Ib Study of Palbociclib plus Nab-Paclitaxel in Patients with Metastatic Adenocarcinoma of the Pancreas. Cancer Res Commun. 2022 Nov 2;2(11):1326-1333. doi: 10.1158/2767-9764.CRC-22-0072. eCollection 2022 Nov. PMID 36970055
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481059&StudyName=An%20Open-label%20Phase%20Ib%20Study%20Of%20Palbociclib%20%28oral%20Cdk%204%2F6%20Inhibitor%29%20Plus%20Abraxane%20%28registered%29%20%28nab-paclitaxel%29%20In%20Patients%20With%20Metastatic%20Pancreatic%20Ductal%20Adenocarcinoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a multiple dose, dose escalation study of palbociclib in combination with nab-paclitaxel (nab-P), in sequential cohorts of adult participants.
Groups:
- DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the starting dose level (DL), participants received palbociclib 75 milligrams (mg) daily for 3 weeks of each 28-day cycle and nab-P 100 milligrams per square miter (mg/m^2) weekly for 3 weeks out of each 28-day cycle.
- DL2A Palbociclib 100mg/Nab-Paclitaxel 100mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 2A, participants received palbociclib 100mg daily for 3 weeks of each 28-day cycle and nab-P 100mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 2B, participants received palbociclib 75mg daily for 3 weeks of each 28-day cycle and nab-P 125mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- DL3A Palbociclib 125mg/Nab-Paclitaxel 100 mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 3A, participants received palbociclib 125mg daily for 3 weeks of each 28-day cycle and nab-P 100mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 3B, participants received palbociclib 100mg daily for 3 weeks of each 28-day cycle and nab-P 125mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2: This was the modified dose regimen 1 (MDR1), participants received palbociclib 75mg once daily on Days 1-21 of each 28-day cycle, plus nab-P 125mg/m^2 biweekly in each 28-day cycle.
- MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2: This was the MDR2, participants received palbociclib 75mg continuous dosing, once daily, plus nab-P 100mg/m^2 biweekly in each 28-day cycle.
- MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2: The estimated maximum tolerated dose (MTD) was the DL associated with <33% of 9 participants experiencing a DLT. The MTD was estimated to be palbociclib 100mg once daily on Days 1-21 plus nab-paclitaxel 125mg/m^2 weekly for 3 weeks of a 28-day cycle based on data from the dose escalation cohorts.
Period: Overall Study
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100mg/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100 mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2
Started | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20
Completed (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20
Not completed — Subject Refused Further Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 3 | 0 | 1 | 1 | 0 | 2 | 4
Not completed — Death | 3 | 4 | 4 | 10 | 10 | 11 | 7 | 15

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Groups:
- DL1 Palbociclib 75 mg/Nab-Paclitaxel 100 mg /m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the starting dose level (DL), participants received palbociclib 75mg daily for 3 weeks of each 28-day cycle and nab-paclitaxel 100mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | DL1 Palbociclib 75 mg/Nab-Paclitaxel 100 mg /m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100mg/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100 mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Total
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 76
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 4
  45-64 | 2 | 5 | 3 | 5 | 6 | 7 | 8 | 9 | 45
  65-75 | 1 | 1 | 1 | 5 | 5 | 4 | 1 | 9 | 27
  >75 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 1 | 6 | 5 | 3 | 6 | 6 | 34
  Male | 1 | 2 | 3 | 5 | 6 | 8 | 3 | 14 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 6 | 4 | 11 | 11 | 11 | 8 | 20 | 74
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Adverse events (AEs) considered as dose limiting toxicities (DLTs) included: hematologic: Grade 4 neutropenia lasting >4 days; Febrile neutropenia (defined as neutropenia Grade>=3 [absolute neutrophil count {ANC}<1000 cells/cubic millimeter {mm^3}] and a body temperature >=38.5 [degrees centigrade]℃) requiring antibiotic or antifungal treatment; any Grade 4 thrombocytopenia (<25000/mm^3 or 25.0*10^9/[liter]L). Non-hematologic: Grade >=3 toxicities, except those that had not been maximally treated (eg, nausea, vomiting, diarrhea). Any AE that caused a palbociclib treatment interruption of greater than 7 consecutive days or caused any combination of interruption/reduction for >=14 days. Any AE that caused omission or reduction of at least 2 of the 3 weekly doses of nab-P.
Time Frame: From Day 1 until pre-dose Cycle 2 Day 1
Population: The analysis population included all participants who received at least 1 dose of either investigational product and met the measurable criteria.
Measure: Count of Participants; unit: Participants
Groups:
- DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 2A, participants received palbociclib 100mg daily for 3 weeks of each 28-day cycle and nab-P 100mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 3A, participants received palbociclib 125mg daily for 3 weeks of each 28-day cycle and nab-P 100mg/m2 weekly for 3 weeks out of each 28-day cycle.
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 6
Participants | 0 | 1 | 0 | 0 | 1 | 1 | 1

2. Secondary Outcome: Number of Participants With Adverse Events
Description: An AE was any untoward medical occurrence in a clinical investigation patient administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An serious AE (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of investigational product. Disease progression was not considered a treatment emergent AE unless the participant died of disease prior to 28 days after discontinuation of treatment. Treatment emergent AEs with cause possibly, probably or definitely related to treatment, as judged by the investigator, were defined as treatment-related AEs. AEs were graded by investigator according to CTCAE v4.03.
Time Frame: From the signing of informed consent up to 56 days after the last administration of the investigational product, or 365 days from the first dose of investigational product, whichever is later
Population: The analysis population included all participants who received at least 1 dose of either investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- MTD+DL3B: The combined DL3B+MTD cohort was 7 first line participants from the DL3B cohort and all participants from the MTD cohort.
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 27
Participants
  All causality treatment-emergent AEs | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 27
  Treatment-related treatment-emergent AEs | 3 | 7 | 4 | 10 | 11 | 11 | 9 | 20 | 27
  All causality SAEs | 2 | 4 | 3 | 4 | 6 | 9 | 2 | 12 | 15
  Treatment-related SAES | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 6 | 6
  All causality Grade 3 or 4 AEs | 3 | 6 | 3 | 9 | 11 | 10 | 5 | 20 | 27
  Treatment-related Grade 3 or 4 AEs | 2 | 5 | 2 | 8 | 11 | 7 | 4 | 20 | 27
  All causality Grade 5 AEs | 0 | 1 | 1 | 1 | 3 | 5 | 0 | 1 | 2
  Treatment-related Grade 5 AEs | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: The number of participants with following laboratory abnormalities meeting any of the Grades 1 to 4 classified according to NCI CTCAE v4.0 were summarized: hematology (anemia, hemoglobin increased, lymphocyte count increased, lymphopenia, neutrophils, platelets and white blood cells) and chemistry laboratory tests (alanine aminotransferase, alkaline phosphatase, amylase, aspartate aminotransferase, bilirubin, creatinine, hypercalcemia, hyperglocemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia, lipase).
Time Frame: From screening to the end of treatment/withdrawal visit (up to 63 days from last dose of investigational product).
Population: The analysis population included all participants who received at least 1 dose of either investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 27
Participants
  Anemia | 3 | 7 | 4 | 11 | 11 | 11 | 8 | 20 | 27
  Hemoglobin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Lymphocyte count increased | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphopenia | 3 | 7 | 2 | 9 | 10 | 11 | 7 | 20 | 27
  Neutrophils (absolute) | 3 | 7 | 2 | 10 | 10 | 9 | 8 | 20 | 27
  Platelets | 2 | 4 | 0 | 8 | 8 | 5 | 1 | 10 | 15
  White blood cells | 3 | 7 | 3 | 10 | 10 | 9 | 8 | 20 | 27
  Alanine aminotransferase (ALT) | 2 | 4 | 1 | 3 | 4 | 4 | 5 | 11 | 15
  Alkaline phosphatase | 2 | 6 | 3 | 9 | 8 | 8 | 6 | 15 | 20
  Amylase: number analyzed (Participants) | 3 | 6 | 3 | 10 | 11 | 10 | 9 | 19 | 26
  Amylase | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2
  Aspartate aminotransferase (AST) | 2 | 3 | 1 | 5 | 6 | 5 | 6 | 8 | 13
  Bilirubin (total) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 4 | 4
  Creatinine | 3 | 7 | 3 | 10 | 11 | 10 | 9 | 18 | 25
  Hypercalcemia | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2
  Hyperglycemia | 3 | 7 | 3 | 9 | 7 | 10 | 7 | 16 | 23
  Hyperkalemia | 0 | 0 | 2 | 1 | 4 | 2 | 3 | 6 | 9
  Hypermagnesemia: number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 10 | 9 | 20 | 27
  Hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Hypernatremia | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 2
  Hypoalbuminemia | 2 | 2 | 3 | 5 | 5 | 7 | 4 | 10 | 13
  Hypocalcemia | 2 | 2 | 2 | 5 | 5 | 5 | 5 | 9 | 12
  Hypoglycemia | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 3 | 6
  Hypokalemia | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 5 | 6
  Hypomagnesemia: number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 10 | 9 | 20 | 27
  Hypomagnesemia | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 3 | 6
  Hyponatremia | 3 | 2 | 3 | 6 | 3 | 3 | 2 | 6 | 8
  Hypophosphatemia: number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 10 | 9 | 20 | 27
  Hypophosphatemia | 0 | 1 | 1 | 4 | 0 | 3 | 2 | 6 | 6
  Liapase: number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 10 | 9 | 20 | 27
  Liapase | 1 | 1 | 1 | 2 | 2 | 2 | 2 | 5 | 6

4. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-specified Criteria
Description: Vital signs evaluation included sitting diastolic blood pressure (DBP), systolic blood pressure (SBP), and pulse rate. Suggest text: Vital signs categorical summary included: 1)SBP>150mmHg or DBP>100mmHg; 2)SBP>200mmHg or DBP>110mmHg; 3)SBP increase >=20 and <40mmHg; 4)SBP increase >=40 and <60mmHg; 5)SBP increase>=60mmHg; 6)DBP increase >=10 and <20mmHg; 7)DBP increase >=20 and <30mmHg; 8)DBP increase >=30mmHg; 9)pulse rate>120bpm; 10)pulse rate<50bpm.
Time Frame: From screening to the end of treatment/withdrawal visit (up to 63 days from last dose of investigational product).
Population: The analysis population included all participants who received at least 1 dose of either investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 27
Participants
  Maximum on-study SBP>150 or DBP>100 | 1 | 1 | 0 | 2 | 2 | 2 | 1 | 4 | 5
  Maximum on-study SBP >200 or DBP>110 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum increase from Baseline SBP>=20 and SBP<40 | 0 | 0 | 0 | 5 | 0 | 2 | 1 | 4 | 4
  Maximum increase from Baseline SBP>=40 and SBP<60 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 3
  Maximum increase from Baseline SBP>=60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum increase from Baseline DBP>=10 and DPB<20 | 0 | 0 | 1 | 3 | 5 | 1 | 4 | 6 | 9
  Maximum increase from Baseline DBP>= 20 and DBP<30 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Maximum increase from Baseline DBP >=30 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Maximum on-study pulse rate (bpm) >120 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum on-study pulse rate (bpm) <50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With 20% Maximum Reduction From Baseline in Ca19-9
Description: Carbohydrate antigen 19-9 (Ca19-9) is a clinical pharmacodynamic (PD) marker associated with metastatic pancreatic ductal adenocarcinoma (mPDAC).
Time Frame: From screening to the end of treatment/withdrawal visit (up to 63 days from last dose of investigational product).
Population: The analysis population included all participants who received at least 1 dose of investigational product and had at least 1 baseline biomarker assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 3 | 8 | 9 | 7 | 6 | 14 | 21
Participants | 3 | 5 | 0 | 7 | 6 | 5 | 3 | 10 | 15

6. Secondary Outcome: Number of Participants With 50% Maximum Reduction From Baseline in Ca19-9
Description: Ca19-9 is a clinical PD marker associated with metastatic mPDAC.
Time Frame: From screening to the end of treatment/withdrawal visit (up to 63 days from last dose of investigational product).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 3 | 8 | 9 | 7 | 6 | 14 | 21
Participants | 1 | 4 | 0 | 5 | 6 | 4 | 2 | 5 | 10

7. Secondary Outcome: Number of Participants With 70% Maximum Reduction From Baseline in Ca19-9
Description: Ca19-9 is a clinical PD marker associated with metastatic mPDAC.
Time Frame: From screening to the end of treatment/withdrawal visit (up to 63 days from last dose of investigational product).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 3 | 8 | 9 | 7 | 6 | 14 | 21
Participants | 0 | 1 | 0 | 3 | 4 | 1 | 1 | 4 | 8

8. Secondary Outcome: Number of Participants With 90% Maximum Reduction From Baseline in Ca19-9
Description: Ca19-9 is a clinical PD marker associated with metastatic mPDAC.
Time Frame: From screening to the end of treatment/withdrawal visit (up to 63 days from last dose of investigational product).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 3 | 8 | 9 | 7 | 6 | 14 | 21
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2

9. Secondary Outcome: Objective Response Rate
Description: Percentage of participants who achieved objective response (OR) based on investigator assessment is presented. OR is defined as a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Objective response rate (ORR) was defined as the percentage of participants with a best overall response of CR or PR relative to all anti-tumor evaluable participants.
Time Frame: From screening to 365 days from the last dose of investigational product
Population: The analysis population included all participants who received at least 1 dose of either investigational product, had a baseline tumor assessment and at least 1 on-treatment tumor assessment prior to any new anti-cancer therapies. Results for groups with a small sample size should be interpreted with caution.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 16 | 23
Percentage of participants |  |  |  |  | 28.6 [3.7 to 71.0] |  |  | 6.3 [0.2 to 30.2] | 13.0 [2.8 to 33.6]

10. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurred first. Disease progression was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm.
Time Frame: From screening to 365 days from the last dose of investigational product
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 16 | 23
Months |  |  |  |  | NA [3.8 to NA] — Number of participants with CR/PR was too small. |  |  | 7.4 [NA to NA] — Number of participants with CR/PR was too small. | 7.4 [3.8 to NA] — Number of participants with CR/PR was too small.

11. Secondary Outcome: Progression Free Survival
Description: The progression free survival (PFS) was defined as the time from the date of first dose to the date of the first documentation of objective tumor progression as per RECIST v1.1 or death due to any cause in the absence of documented progression disease, whichever occurred first.
Time Frame: From screening to 365 days from the last dose of investigational product
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 27
Months | 9.1 [3.7 to 9.1] | 9.5 [1.8 to NA] — Since not all participants had disease progression, the upper bound 95% CI cannot be estimated. | 1.7 [1.4 to 1.9] | 3.5 [1.7 to 7.2] | 5.5 [0.8 to 14.5] | 5.3 [1.6 to 6.9] | 1.8 [1.5 to 8.6] | 3.8 [2.4 to 9.7] | 5.3 [3.5 to 9.7]

12. Secondary Outcome: Six-month Progression-free Survival Rate (6m-PFSR)
Description: 6m-PFS was defined as PFS status (progression free and alive, or not) at Month 6. It was summarized as a product limit estimator based on the Kaplan-Meier method to account for censored events.
Time Frame: From screening to 6 months after first dose of investigational product
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 27
Percentage of participants | 66.7 [5.4 to 94.5] | 66.7 [19.5 to 90.4] | NA [NA to NA] — Since not all participants had disease progression, 6m-PFSR and associated 95% CI cannot be estimated. | 30.0 [7.1 to 57.8] | 36.4 [11.2 to 62.7] | 27.3 [6.5 to 53.9] | 25.0 [3.7 to 55.8] | 36.2 [13.4 to 59.9] | 36.5 [17.0 to 56.3]

13. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose to the date of death due to any cause. Following the end of treatment visit, survival status was collected in all participants every month until 12 months (365 days) had elapsed from the last dose of investigational product.
Time Frame: From screening to 365 days from the last dose of investigational product
Population: Participants who received study treatment, had adequate baseline assessments and at least 1 on-treatment tumor assessment prior to any new anti-cancer therapies were evaluable for anti-tumor activity. Results for groups with a small sample size should be interpreted with caution.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 27
Months | 9.8 [8.8 to 16.3] | 23.4 [5.6 to NA] — Four (4) participants died and 3 were censored. | 3.3 [2.1 to 7.7] | 7.2 [4.0 to 15.3] | 9.9 [0.8 to 14.8] | 5.3 [2.4 to 11.7] | 7.2 [4.0 to NA] — Seven (7) participants died and 2 were censored. | 11.4 [4.5 to 14.9] | 12.1 [6.4 to 14.8]

14. Secondary Outcome: Number of Participants With Positive p16
Description: p16 is a tumor suppressor protein which plays an important role in cell cycle regulation. The analysis of biomarker p16 expression might aid in the identification of patient subpopulations most likely to benefit from treatment. The results from p16 expression testing by immunohistochemistry (IHC) was used for sensitivity analyses. (a) and (b) :p16 cutoff utilizing the optimal cut point identified by the ORC analysis for the OS (a) or PFS (b) and the p16 positive tumor cells.
Time Frame: From Day-2 to up to 63 days from last dose of investigational product
Population: The analysis population included all participants who received at least 1 dose of investigational product and had at least 1 baseline biomarker assessment and met the criteria for measuring p16.
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 5 | 4 | 10 | 10 | 10 | 9 | 19 | 26
Participants
  p16(a) | 1 | 2 | 0 | 5 | 7 | 6 | 3 | 10 | 15
  p16(b) | 1 | 1 | 0 | 4 | 6 | 4 | 1 | 9 | 13

15. Secondary Outcome: Retinoblastoma Protein (Rb) Percent Positive Cell (Nuclear Staining)
Description: Rb is a tumor suppressor protein that is dysfunctional in several major cancers. The results from Rb expression testing by IHC was used for sensitivity analyses.
Time Frame: From Day-2 to up to 63 days from last dose of investigational product
Population: The analysis population included all participants who received at least 1 dose of investigational product and had at least 1 baseline biomarker assessment and met the criteria for measuring Rb.
Measure: Mean (Standard Deviation); unit: Percentage of positive cell
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 5 | 4 | 10 | 10 | 10 | 9 | 19 | 26
Percentage of positive cell | 88.3 (7.64) | 80.0 (29.79) | 68.8 (23.23) | 91.1 (10.24) | 90.5 (18.77) | 92.5 (8.25) | 82.2 (32.70) | 92.4 (19.10) | 91.7 (19.54)

16. Secondary Outcome: Rb H-score Nuclear Staining
Description: Rb is a tumor suppressor protein that is dysfunctional in several major cancers. The results from Rb expression testing by IHC was used for sensitivity analyses. The H-score is a method of assessing the extent of nuclear immunoreactivity, applicable to steroid receptors. The score is obtained by the formula: 3*percentage of strongly staining nuclei + 2*percentage of moderately staining nuclei + percentage of weakly staining nuclei, giving the range of 0 to 300
Time Frame: From Day-2 to up to 63 days from last dose of investigational product
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
Number analyzed (Participants) | 3 | 5 | 4 | 10 | 10 | 10 | 9 | 19 | 26
Scores on a scale | 158.3 (34.03) | 154.0 (65.9) | 108.8 (43.28) | 166.7 (32.88) | 176.0 (47.31) | 172.5 (32.17) | 145.6 (70.51) | 187.9 (52.37) | 185.4 (51.63)

17. Secondary Outcome: Palbociclib Multiple Dose Maximum Plasma Concentration (Cmax)
Description: The palbociclib multiple dose maximum plasma concentration(Cmax) was observed directly from data.
Time Frame: Cycle 1 Day 13 at 0 (pre-dose), 2, 4, 6, 8 and 24 hours post palbociclib dose, and pre-dose on Cycle 2, Days 1 and 15.
Population: The analysis population included all enrolled participants treated who had sufficient information to estimate at least 1 of the pharmacokinetic (PK) of interest and had no major protocol deviations affecting PK assessment. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milli liter (ng/mL)
Groups:
- Overall Participants With Dose Normalized to 125 mg/m^2: The overall participants with dose normalized to 125 mg/m^2
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2
Number analyzed (Participants) | 2 | 6 | 3 | 6 | 7 | 10 | 8 | 15 | 57
nanogram per milli liter (ng/mL) | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 90.68 (24) | 57.30 (56) | 98.79 (46) | 64.55 (23) | 48.05 (54) | 53.65 (25) | 70.14 (43) | 90.44 (39)

18. Secondary Outcome: Palbociclib Multiple Dose Time for Cmax (Tmax)
Description: The palbociclib multiple dose time for Cmax (Tmax) was observed directly from data.
Time Frame: Cycle 1 Day 13 at 0 (pre-dose), 2, 4, 6, 8 and 24 hours post palbociclib dose, and pre-dose on Cycle 2, Days 1 and 15.
Population: as for outcome 17
Measure: Median (Full Range); unit: hour(hr)
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 2 | 6 | 3 | 6 | 7 | 10 | 8 | 15 | 57
hour(hr) | 4.93 [4.20 to 5.65] | 5.00 [4.00 to 7.92] | 3.90 [3.00 to 24.0] | 5.83 [4.05 to 25.0] | 4.50 [3.88 to 6.25] | 5.00 [1.83 to 7.17] | 6.01 [0 to 8.00] | 4.17 [0.600 to 7.98] | 5.05 [0 to 25.0]

19. Secondary Outcome: Palbociclib Area Under the Plasma Concentration-time Curve for Dosing Interval τ (AUCτ)
Description: The palbociclib area under the plasma concentration-time curve for dosing interval τ (AUCτ) was observed directly from data.
Time Frame: Cycle 1 Day 13 at 0 (pre-dose), 2, 4, 6, 8 and 24 hours post palbociclib dose, and pre-dose on Cycle 2, Days 1 and 15.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milli liter (ng.hr/mL)
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 2 | 6 | 3 | 6 | 7 | 10 | 8 | 15 | 57
nanogram*hour per milli liter (ng.hr/mL) | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 1497 (18) | 897.4 (36) | 1867 (40) | 1169 (21) | 767.9 (42) | 967.7 (26) | 1251 (38) | 1569 (34)

20. Secondary Outcome: Palbociclib Multiple Dose Trough Plasma Concentration(Ctrough)
Description: The palbociclib multiple dose trough plasma concentration (Ctrough) was observed directly from data.
Time Frame: Cycle 1 Day 13 at 0 (pre-dose), 2, 4, 6, 8 and 24 hours post palbociclib dose, and pre-dose on Cycle 2, Days 1 and 15.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 2 | 6 | 3 | 6 | 6 | 10 | 8 | 15 | 56
ng/mL | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 43.42 (34) | 26.84 (19) | 71.82 (42) | 41.92 (11) | 22.34 (37) | 30.66 (34) | 34.89 (34) | 48.51 (38)

21. Secondary Outcome: Palbociclib Multiple Dose Apparent Clearance (CL/F)
Description: The palbociclib multiple dose apparent clearance (CL/F) was observed directly from data.
Time Frame: Cycle 1 Day 13 at 0 (pre-dose), 2, 4, 6, 8 and 24 hours post palbociclib dose, and pre-dose on Cycle 2, Days 1 and 15.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 2 | 6 | 3 | 6 | 7 | 10 | 8 | 15 | 57
liter per hour (L/hr) | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 66.67 (18) | 83.63 (36) | 64.52 (40) | 85.42 (21) | 97.67 (42) | 77.62 (26) | 79.95 (38) | 79.35 (34)

22. Secondary Outcome: Nab-P Cmax
Description: The nab-P Cmax on Cycle 1 Day -1 and Day 13 were observed directly from data.
Time Frame: Prior to nab-P infusion and at 30 min (end of infusion), 1, 2, 4, 6, 8, 24, and 48 hours post the start of paclitaxel infusion on Day -2 and 13 of Cycle 1.
Population: The analysis population included all enrolled participants treated who were treated. Number analyzed for each category represents the number of participants with Nab-P Cmax data for each time point. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 3 | 7 | 3 | 11 | 11 | 11 | 8 | 19 | 76
ng/mL
  Day -1: number analyzed (Participants) | 3 | 7 | 3 | 11 | 11 | 11 | 8 | 19 | 73
  Day -1 | 1208 (250) | 1595 (61) | 1869 (47) | 2733 (127) | 3396 (117) | 3271 (113) | 1851 (196) | 3054 (129) | 2827 (121)
  Day 13: number analyzed (Participants) | 2 | 6 | 3 | 7 | 7 | 10 | 8 | 15 | 58
  Day 13 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 1532 (146) | 2316 (56) | 1265 (219) | 3073 (57) | 2821 (93) | 1266 (167) | 3448 (73) | 2487 (111)

23. Secondary Outcome: Nab-P Tmax
Description: The nab-P Tmax on Day -1 and Day 13 were observed directly from data.
Time Frame: as for outcome 22
Population: The analysis population included all enrolled participants treated who were treated. Number analyzed for each category represents the number of participants with Nab-P Tmax data for each time point. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Median (Full Range); unit: hr
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 76
hr
  Day -1: number analyzed (Participants) | 3 | 7 | 3 | 11 | 11 | 11 | 8 | 19 | 73
  Day -1 | 0.500 [0.500 to 1.00] | 1.00 [0.500 to 1.13] | 1.00 [0.517 to 1.00] | 0.567 [0.483 to 1.00] | 0.600 [0.483 to 1.00] | 0.500 [0.450 to 1.03] | 0.775 [0.500 to 1.00] | 0.500 [0.000 to 1.17] | 0.517 [0.000 to 1.17]
  Day 13: number analyzed (Participants) | 2 | 6 | 3 | 7 | 7 | 10 | 8 | 15 | 58
  Day 13 | 0.592 [0.583 to 0.600] | 0.583 [0.500 to 1.20] | 0.500 [0.500 to 1.00] | 1.00 [0.500 to 1.05] | 0.517 [0.467 to 1.00] | 0.500 [0.450 to 1.17] | 0.575 [0.500 to 1.03] | 0.533 [0.467 to 1.50] | 0.542 [0.450 to 1.50]

24. Secondary Outcome: Nab-P Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration (AUClast)
Description: The nab-P area under the plasma concentration-time curve from time 0 to last quantifiable concentration (AUClast) on Day -1 and Day 13 were observed directly from data.
Time Frame: as for outcome 22
Population: The analysis population included all enrolled participants treated who were treated. Number analyzed for each category represents the number of participants with Nab-P AUClast data for each time point. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 76
ng.hr/mL
  Day -1: number analyzed (Participants) | 3 | 7 | 3 | 11 | 11 | 11 | 8 | 19 | 73
  Day -1 | 2071 (127) | 3501 (48) | 3489 (33) | 4291 (70) | 4895 (54) | 4472 (59) | 2632 (146) | 3942 (60) | 4211 (70)
  Day 13: number analyzed (Participants) | 2 | 5 | 3 | 7 | 7 | 10 | 8 | 15 | 57
  Day 13 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 2592 (70) | 4096 (64) | 2894 (133) | 4095 (32) | 4183 (44) | 2071 (100) | 4269 (52) | 3812 (67)

25. Secondary Outcome: Nab-P Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinite Time (AUCinf)
Description: The nab-P area under the plasma concentration-time curve from time 0 extrapolated to infinite time (AUCinf) on Day -1 and Day 13 observed directly from data.
Time Frame: as for outcome 22
Population: The analysis population included all enrolled participants treated who were treated. Number analyzed for each category represents the number of participants with Nab-P AUCinf data for each time point. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 76
ng.hr/mL
  Day -1: number analyzed (Participants) | 2 | 7 | 3 | 10 | 10 | 9 | 7 | 14 | 62
  Day -1 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 3851 (50) | 3780 (30) | 4157 (48) | 5387 (54) | 5132 (56) | 4116 (34) | 4760 (49) | 4977 (46)
  Day 13: number analyzed (Participants) | 2 | 2 | 3 | 3 | 7 | 9 | 6 | 13 | 45
  Day 13 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 4590 (60) | 3349 (67) | 4493 (29) | 4482 (46) | 2206 (118) | 5135 (38) | 4447 (55)

26. Secondary Outcome: Nab-P Terminal Plasma Elimination Half-life (t1/2)
Description: The nab-P t1/2 on Day -1 and Day 13 were observed directly from data.
Time Frame: as for outcome 22
Population: The analysis population included all enrolled participants treated who were treated. Number analyzed for each category represents the number of participants with Nab-P t1/2 data for each time point. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Median (Full Range); unit: hr
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 76
hr
  Day -1: number analyzed (Participants) | 2 | 7 | 3 | 10 | 10 | 9 | 7 | 14 | 62
  Day -1 | 16.95 [16.6 to 17.3] | 11.10 [7.75 to 18.6] | 12.00 [10.9 to 16.6] | 15.25 [10.0 to 20.1] | 12.85 [9.41 to 16.1] | 16.10 [9.30 to 31.3] | 15.80 [9.31 to 20.4] | 14.45 [8.86 to 20.8] | 14.50 [7.75 to 31.3]
  Day 13: number analyzed (Participants) | 2 | 2 | 3 | 3 | 7 | 9 | 6 | 13 | 45
  Day 13 | 15.20 [13.4 to 17.0] | 17.65 [13.0 to 22.3] | 18.60 [12.3 to 20.8] | 16.40 [15.7 to 19.3] | 17.10 [7.51 to 21.9] | 13.80 [9.82 to 18.8] | 14.35 [2.76 to 18.8] | 14.40 [9.26 to 24.3] | 15.20 [2.76 to 24.3]

27. Secondary Outcome: Nab-P Clearance (CL)
Description: The nab-P clearance on Day -1 and Day 13 were observed directly from data.
Time Frame: as for outcome 22
Population: The analysis population included all enrolled participants treated who were treated. Number analyzed for each category represents the number of participants with Nab-P clearance data for each time point. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 76
liter per hour (L/hr)
  Day -1: number analyzed (Participants) | 2 | 7 | 3 | 10 | 10 | 9 | 7 | 14 | 62
  Day -1 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 42.05 (56) | 60.94 (36) | 41.69 (51) | 37.77 (46) | 44.02 (51) | 42.39 (34) | 47.39 (48) | 43.63 (46)
  Day 13: number analyzed (Participants) | 2 | 2 | 3 | 3 | 7 | 9 | 6 | 13 | 45
  Day 13 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 52.34 (65) | 50.14 (78) | 46.37 (33) | 47.89 (48) | 76.34 (131) | 44.92 (40) | 49.35 (57)

28. Secondary Outcome: Nab-P Volume of Distribution (Vz)
Description: The nab-P on Day -1 and Day 13 were observed directly from data.
Time Frame: as for outcome 22
Population: The analysis population included all enrolled participants treated who were treated. Number analyzed for each category represents the number of participants with Nab-P volume of distribution data for each time point. Results for groups with a small sample size could be misleading due to inter-individual variability and should be interpreted with caution.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | DL1 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg/Nab-Paclitaxel 100/m^2 | DL2B Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg/Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | Overall Participants With Dose Normalized to 125 mg/m^2.
Number analyzed (Participants) | 3 | 7 | 4 | 11 | 11 | 11 | 9 | 20 | 76
L
  Day -1: number analyzed (Participants) | 2 | 7 | 3 | 10 | 10 | 9 | 7 | 14 | 62
  Day -1 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 709.1 (44) | 1140 (44) | 891.3 (37) | 701.6 (46) | 943.3 (56) | 904.5 (39) | 950.8 (51) | 873.3 (46)
  Day 13: number analyzed (Participants) | 2 | 2 | 3 | 3 | 7 | 9 | 6 | 13 | 45
  Day 13 | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | NA (NA) — It is Pfizer convention that the geometric mean value and CV% to be calculated from at least 3 data points, the number of participants was insufficient. | 1271 (106) | 1235 (69) | 1070 (71) | 927.2 (32) | 1220 (57) | 971.1 (52) | 1036 (52)

ADVERSE EVENTS:
Time Frame: From the signing of informed consent up to 56 days after the last administration of the investigational product, or 365 days from the first dose of investigational product, whichever is later.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Groups:
- DL1 Palbociclib 75mg / Nab-Paclitaxel 100mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the starting dose level (DL), participants received palbociclib 75 milligrams (mg) daily for 3 weeks of each 28-day cycle and nab-P 100 milligrams per square miter (mg/m^2) weekly for 3 weeks out of each 28-day cycle.
- DL2A Palbociclib 100mg / Nab-Paclitaxel 100mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 2A, participants received palbociclib 100mg daily for 3 weeks of each 28-day cycle and nab-P 100mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- DL2B Palbociclib 75mg / Nab-Paclitaxel 125mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 2B, participants received palbociclib 75mg daily for 3 weeks of each 28-day cycle and nab-P 125mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- DL3A Palbociclib 125mg / Nab-Paclitaxel 100mg/m^2: Consecutive cohorts of participants received escalating doses of oral palbociclib in combination with intravenous nab-P in 28-day cycles. This was the escalated DL 3A, participants received palbociclib 125mg daily for 3 weeks of each 28-day cycle and nab-P 100mg/m^2 weekly for 3 weeks out of each 28-day cycle.
- MTD+DL3B: The combined DL3B+MTD cohort was 7 first line participants from the DL3B cohort and all patients from the MTD cohort.
Arm/Group | DL1 Palbociclib 75mg / Nab-Paclitaxel 100mg/m^2 | DL2A Palbociclib 100mg / Nab-Paclitaxel 100mg/m^2 | DL2B Palbociclib 75mg / Nab-Paclitaxel 125mg/m^2 | DL3A Palbociclib 125mg / Nab-Paclitaxel 100mg/m^2 | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 | MTD+DL3B
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/7 | 3/4 | 2/11 | 3/11 | 5/11 | 2/9 | 6/20 | 7/27
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/7 | 3/4 | 4/11 | 6/11 | 9/11 | 2/9 | 12/20 | 15/27
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 4/4 | 11/11 | 10/11 | 11/11 | 9/9 | 20/20 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL1 Palbociclib 75mg / Nab-Paclitaxel 100mg/m^2 (N=3) | DL2A Palbociclib 100mg / Nab-Paclitaxel 100mg/m^2 (N=7) | DL2B Palbociclib 75mg / Nab-Paclitaxel 125mg/m^2 (N=4) | DL3A Palbociclib 125mg / Nab-Paclitaxel 100mg/m^2 (N=11) | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 (N=11) | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 (N=11) | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 (N=9) | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 (N=20) | MTD+DL3B (N=27)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstrucion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL1 Palbociclib 75mg / Nab-Paclitaxel 100mg/m^2 (N=3) | DL2A Palbociclib 100mg / Nab-Paclitaxel 100mg/m^2 (N=7) | DL2B Palbociclib 75mg / Nab-Paclitaxel 125mg/m^2 (N=4) | DL3A Palbociclib 125mg / Nab-Paclitaxel 100mg/m^2 (N=11) | DL3B Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 (N=11) | MDR1 Palbociclib 75mg/Nab-Paclitaxel 125mg/m^2 (N=11) | MDR2 Palbociclib 75mg/Nab-Paclitaxel 100mg/m^2 (N=9) | MTD Palbociclib 100mg/Nab-Paclitaxel 125mg/m^2 (N=20) | MTD+DL3B (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (5) | 2 (3) | 5 (11) | 3 (6) | 6 (11) | 1 (1) | 9 (17) | 11 (22)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (10) | 0 (0) | 2 (6) | 0 (0) | 2 (3) | 2 (5) | 2 (11) | 2 (11)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (6) | 5 (37) | 1 (2) | 9 (57) | 7 (21) | 5 (10) | 6 (19) | 16 (63) | 20 (78)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (6) | 1 (1) | 0 (0) | 5 (12) | 6 (18)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (6) | 0 (0) | 1 (1) | 2 (5) | 4 (9) | 5 (5) | 4 (6) | 5 (9)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 2 (2) | 3 (4) | 1 (1) | 7 (8) | 8 (9)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (13) | 1 (1) | 2 (5) | 4 (6) | 5 (11) | 2 (3) | 9 (17) | 12 (22)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (7) | 1 (1) | 4 (5) | 5 (8) | 6 (9) | 4 (10) | 9 (12) | 13 (19)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (2) | 1 (1) | 1 (1) | 6 (13) | 5 (7) | 3 (3) | 4 (6) | 9 (16)
Asthenia (General disorders) | 1 (1) | 3 (11) | 1 (2) | 2 (6) | 3 (14) | 4 (6) | 2 (9) | 4 (18) | 7 (32)
Catheter site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Early satiety (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 3 (7) | 2 (2) | 7 (9) | 9 (12)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 2 (4)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 4 (10) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 5 (9) | 6 (10)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deficiency of bile secretion (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perinephric abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (2) | 1 (2)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (2) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (7) | 5 (9)
Neutrophil count decreased (Investigations) | 1 (2) | 2 (6) | 0 (0) | 1 (4) | 2 (10) | 0 (0) | 0 (0) | 1 (2) | 3 (12)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 4 (8) | 2 (3) | 2 (5) | 2 (4) | 5 (6) | 7 (9)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 2 (6) | 1 (2) | 1 (1) | 4 (10) | 7 (14) | 5 (9) | 3 (8) | 7 (18)
Dehydration (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (5) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (15) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 1 (3) | 1 (1) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 4 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (5) | 1 (2) | 0 (0) | 4 (6) | 6 (11)
Neurotoxicity (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 4 (11) | 6 (15)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Semnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Confusion state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choluria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 3 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 3 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (6) | 1 (1) | 3 (3) | 4 (5) | 6 (10) | 3 (3) | 6 (8) | 9 (12)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 5 (5)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 2 (4) | 2 (4)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The rationale for the study was supported on theoretical and preclinical grounds. However, based on emerging clinical data, the combination of palbociclib and nab-P was not to be further developed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02501902/SAP_000.pdf
  • Study Protocol (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT02501902/Prot_001.pdf